CLINICAL TRIAL: NCT06639126
Title: Intervention Study Focused on the Intestinal Microbiome to Evaluate the Impact of a Wild Thyme Extract (Thymus Serpyllum) Extract With Anti-inflammatory and Metabolic Properties Against Functional Gastrointestinal Disorders.
Acronym: InT-FGD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental (Other)
Responsible Party: Principal Investigator, Alba Rodriguez Nogales, Professor, Advanced Bionics
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FIBAO-UGR
Record Dates: First submitted 2024-09-20; First posted 2024-10-15 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-10

CONDITIONS: Functional Gastrointestinal Disorders
Keywords: Intestinal microbiota; Functional dyspepsia; Thymus vulgaris; Functional gastrointestinal disorders
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — microcrystalline cellulose; thyme extract

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo treated with 600 mg/capsule/day of microcrystalline cellulose
  Interventions: Other: Placebo
- Active (Experimental): Group with wild thyme extract
  Interventions: Dietary Supplement: Wild thyme extract

INTERVENTIONS:
Dietary Supplement: Wild thyme extract — All patients will be randomized (1:1) to receive the active thyme extract (600 mg/capsule/day or 600 mg/capsule/day of microcrystalline cellulose) in the form of capsules, administered orally and daily for 2 months
  Other Names: 600 mg/capsule/day of microcrystalline cellulose; 600 mg/capsule/day of thyme extract
  Arms: Active
Other: Placebo — 600 mg/day microcrystalline cellulose
  Arms: Placebo

SUMMARY:
Functional gastrointestinal disorders (FGD), now known as disorders of gut-brain interactions (DGBI), are characterized by gastrointestinal symptoms linked to motility issues, visceral sensitivity, intestinal permeability, immune activation, neuroendocrine function, CNS processing, and gut microbiota. These disorders include symptoms like abdominal pain, diarrhea, constipation, bloating, fullness, nausea, and vomiting, associated with conditions like IBS and functional dyspepsia. The complex pathophysiology of FGDs is not fully understood, affecting one-third of gastroenterology consultations. Diagnosis and treatment follow Rome Foundation criteria, focusing on symptom management rather than underlying mechanisms. Nearly half the population will meet FGD criteria at some point, with significant overlap in symptoms and conditions.

The gut microbiota's role is crucial, affecting homeostasis and linked to FGDs through dysbiosis. Treatments include antibiotics, dietary changes, and fecal transplants. Prebiotics, including medicinal plant extracts like wild thyme (Thymus serpyllum L.), show promise. Wild thyme has traditionally treated respiratory and gastrointestinal issues and contains phenolic compounds with potential spasmolytic and antioxidant effects.

Preclinical studies show wild thyme extract benefits in inflammation, IBS, and metabolic syndrome models. Recent human trials indicate improvements in gut regularity and microbiota. This study proposes wild thyme extract as a dietary supplement to benefit digestive health in FGDs, hypothesizing its immunomodulatory and prebiotic properties can reduce inflammation and restore microbiota balance. Specific objectives include analyzing microbiome impact, barrier function, inflammation, and identifying prognostic biomarkers to predict treatment response.

DETAILED DESCRIPTION:
Functional gastrointestinal disorders (FGD), recently referred to as disorders of gut-brain interactions (DGBI), are characterized by the presence of gastrointestinal symptoms related to abnormalities in motility, visceral sensitivity, intestinal permeability, immune activation, neuroendocrine function, central nervous system processing, and gut microbiota. The spectrum of symptoms occurring in these FGDs includes abdominal pain, diarrhea, constipation, bloating, a sense of fullness, nausea, and vomiting, and are associated with conditions such as irritable bowel syndrome (IBS), functional dyspepsia, recurrent abdominal pain, or functional constipation/diarrhea, etc. Generally, these diseases are marked by a highly complex pathophysiology that is not fully understood, representing at least one-third of medical consultations related to Gastroenterology. Diagnosis and classification are performed using standardized criteria recommended by the Rome Foundation. Additionally, current treatment approaches target predominant gastrointestinal and psychological symptoms, rather than identifying and addressing specific underlying pathophysiological mechanisms. Nearly half of the general population will meet the criteria for these disorders at some point, and these conditions often overlap within the same individual. IBS is one of the most frequent FGDs, manifesting with recurrent abdominal pain and alterations in stool form and frequency, with a prevalence reaching approximately 4-11% of the population. Functional dyspepsia is characterized by the presence of one or more of the following symptoms: postprandial fullness, early satiety, epigastric pain, or burning, unexplained by routine clinical examination, with a prevalence of around 7%. Functional constipation is associated with difficult, infrequent, or incomplete defecation symptoms that do not meet IBS criteria, and may include abdominal pain with or without bloating, though these symptoms are not predominant, with a prevalence of around 12%. In the case of functional diarrhea, there is recurrent passage of loose, watery stools that do not meet the criteria for IBS, where abdominal pain with or without bloating may be present but is not predominant; the estimated prevalence can reach up to 5%. Another condition that may be included is functional abdominal bloating and distension, characterized by subjective symptoms of abdominal heaviness, pressure, or a feeling of trapped gas (bloating), and an objectively measurable increase in abdominal girth (distension), which do not meet criteria for another functional intestinal disorder (although mild abdominal pain or minor changes in bowel habits may coexist), with a prevalence of around 3%. Finally, up to 11% of FGD cases have been proposed to have intestinal symptoms that cannot be attributed to an organic cause and do not meet the diagnostic criteria for the aforementioned conditions: irritable bowel syndrome, functional constipation, functional diarrhea, with or without bloating. A global survey conducted by the Rome Foundation has established that women have a higher frequency of experiencing some type of FGD (49%) compared to men (37%). Besides gender, several factors seem to increase the risk of developing these digestive disorders: gastroenteritis, a history of trauma or abuse, stress, psychological disorders (anxiety, depression), somatic symptoms (fatigue, headaches, and back pain), obesity, and lack of sleep. Due to the great diversity of diseases that can be considered as FGDs, it is currently not possible to establish a common therapeutic strategy for all of them. In this regard, the general principles of treatment are based on understanding the complexity of the pathophysiology of the disease in question, aiming to improve the dysregulation of the gut-brain axis, which appears to occur frequently. Therefore, the type of symptoms, their location, and physiological determinants will influence the treatment. Some simple and cost-effective treatments, such as laxatives or antidiarrheals, may be sufficient for some patients, although the scientific evidence for these treatments is limited. In the case of functional constipation or IBS with constipation, meta-analysis studies have shown the efficacy of drugs such as linaclotide or lubiprostone (which act as secretagogues through intestinal ion channels), or prokinetics such as prucalopride or tegaserod (which act through serotonin receptors (5-HT)); for diarrhea in IBS, rifaximin (a low-absorption intestinal antibiotic) or alosetron or ondansetron (5-HT3 receptor antagonists) are beneficial. However, if there is severe abdominal pain, treatment may include an antidepressant. Despite the existence of these treatments, not all are effective in all patients, so a significant proportion do not achieve satisfactory therapeutic benefit. Additionally, these treatments are not exempt from the risk of adverse reactions, which may exacerbate the delicate situation presented by some patients. Therefore, the development of new therapeutic strategies for FGDs, combining efficacy and safety, is of great interest for managing these patients. The gut microbiota comprises the set of microorganisms that develop in the intestine, establishing a symbiotic relationship with the host and being involved in numerous functions. Moreover, the gut microbiota communicates with the brain through neural signaling channels (autonomic and enteric nervous systems), endocrine (hypothalamic-pituitary-adrenal axis and enteroendocrine cells), and immune pathways. In fact, several studies have pointed out that the gut-brain microbiota axis is crucial for maintaining homeostasis, and its alteration may be related to the appearance of neurological disorders, thus contributing to the development of other conditions with a significant psychological component, such as FGDs. In this sense, it is currently accepted that the gut microbiota plays an important role in FGDs; supporting this, it has been shown that patients with IBS have a different gastrointestinal microbiome compared to healthy subjects, leading to a situation called intestinal dysbiosis. Furthermore, it has even been proposed that a specific composition of the gut microbiota may influence disease severity. On the other hand, it has also been indicated that alterations in the production of metabolites derived from the metabolic activity of the gut microbiota will actively participate in the development of these diseases. These metabolites include short-chain fatty acids (SCFAs) (acetate, propionate, and butyrate), metabolites derived from amino acids, and bile acids. In line with the above, this dysbiosis situation that seems to characterize various FGDs has led to the development of different treatment approaches aimed at alleviating the symptoms of these diseases, such as IBS, through manipulation of the luminal gut microbiota. Initially, these treatments could include non-absorbable antibiotics (such as rifaximin or neomycin), as well as dietary treatments (low-fermentable oligosaccharide diets, prebiotics, probiotics) and fecal microbiota transplantation. Prebiotics are defined as substrates that will be selectively utilized by microorganisms present in the intestinal lumen, thereby conferring a health benefit to the host. Traditionally, the term prebiotic was restricted to certain dietary carbohydrates; however, it is now accepted that medicinal plant extracts, which can influence the composition of the gut microbiota, may also be considered prebiotics. In this regard, various human studies with medicinal plant extracts have reported their ability to improve symptoms in patients suffering from FGDs. However, most of these trials have used small sample sizes, are observational, and use preparations or formulations that are not commercially available, which constitutes a significant limitation in these studies. Wild thyme (Thymus serpyllum L.) is a perennial shrub native to northern and central Europe. Its aerial parts have been used in Traditional Medicine to treat conditions related to the respiratory and gastrointestinal systems. Regarding the latter, it has been used for the symptomatic treatment of digestive disorders such as epigastric bloating, slow digestion, gas, and flatulence. The presence of non-volatile phenolic compounds, including flavonoids, polyphenolic acids, and triterpenes in these extracts, could justify their spasmolytic effects, as well as the stimulation of gastric juice secretion that facilitates food digestion. Moreover, these active compounds may exert antioxidant properties, making these extracts a potential source of natural antioxidants for the development of nutritional supplements or functional foods in the food industry. Preclinical studies have demonstrated that wild thyme extract has beneficial effects in experimental models of intestinal inflammation and irritable bowel syndrome, as well as in an experimental model of diet-induced metabolic syndrome in mice. In all these cases, the extract improved the chronic inflammatory state associated with the studied experimental models, potentially improving intestinal barrier function and restoring the intestinal dysbiosis characteristic of these intestinal and metabolic diseases. Recently, the first human clinical trial on the impact of a Thymus serpyllum extract formulation has been published, showing benefits in intestinal regularity and gut microbiota. Considering all the above, it is logical to think that the consumption of T. serpylli extract could benefit human digestive health. Therefore, we propose to conduct an intervention study with wild thyme extract as a dietary supplement to corroborate its health benefits against gastrointestinal discomforts, such as FGDs. Consequently, the hypothesis of the present study is related to FGDs being associated with alterations in intestinal homeostasis, where the loss of intestinal barrier function along with a situation of intestinal dysbiosis seem to play a key role in their development. Therefore, the administration of medicinal plant extracts with immunomodulatory and prebiotic properties may exert beneficial effects in these patients, given the lack of an optimal therapeutic strategy that combines efficacy and safety so far. Thus, the hypotheses proposed in this study are: H1: Dietary supplementation with wild thyme extract, with proven immunomodulatory properties, may have beneficial effects on FGDs by reducing the inflammatory response generated in these conditions. H2: Consumption of wild thyme extract in patients with FGDs could positively impact the dysbiosis situation characterizing these disorders by restoring the composition and function of the microbiome. H3: Analysis of the patient's microbiome could act as a predictive biomarker of treatment response. To confirm these hypotheses, the general objective is to analyze the impact of dietary intervention with a well-characterized wild thyme (T. serpylli) extract on the clinical response and prognosis of patients diagnosed with an FGD. With this general objective, several specific objectives are proposed: i) to analyze the impact on the composition of the gut microbiome in patients with FGDs; ii) to determine prognostic biomarkers through the analysis of microbiome parameters to predict clinical response, objective response rate to treatment, and disease progression.

ELIGIBILITY:
Inclusion Criteria:

-Clinical diagnosis of functional gastrointestinal disorder.

Exclusion Criteria:

* Obesity.
* Antibiotic treatment.
* Pregnancy.
* Clinical diagnoses of Inflammatory bowel disease.
* Clinical diagnosis of Celiac disease
* Clinical diagnosis of Hematological pathologies.
* Clinical diagnosis of Autoimmune or immunodeficiency diseases.
* Treatments with opioids, prokinetics, laxatives, antispasmodics, NSAIDs and proton pump inhibitors (PPIs).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the composition of the intestinal microbiome | From enrollment to the end of treatment at 8 weeks
  Metagenomic studies from feces samples at two different points (initial and final point). Shallow shotgun metagenomic will se used to evaluate the composition of the gut microbiota in these samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Alba Rodriguez Nogales, Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruiz-Malagon AJ, Rodriguez-Sanchez MJ, Rodriguez-Sojo MJ, Vezza T, Pischel I, Algieri F, Rodriguez-Cabezas ME, Rodriguez-Nogales A, Galvez J. Intestinal anti-inflammatory and visceral analgesic effects of a Serpylli herba extract in an experimental model of irritable bowel syndrome in rats. Front Pharmacol. 2022 Sep 2;13:967644. doi: 10.3389/fphar.2022.967644. eCollection 2022. PMID 36120292
- [Background] Pavel M, Vostinaru O, Mogosan C, Ghibu S. Phytochemical and pharmacological research on some extracts obtained from Serpylli herba. Farmacia 2011;59:77-84.
- [Background] Knaub, K., Schön, C., Suarez, C.G. and Pischel, I. (2022) Effects of a Food Supplement with a Wild Thyme (Thymus serpyllum L.) Extract on Gut Health and the Microbiome in Humans: A Randomized, Double-Blinded, Placebo-Controlled Clinical Trial. Food and Nutrition Sciences, 2022;13:931-949.
- [Background] Ruiz-Malagon AJ, Rodriguez-Sojo MJ, Hidalgo-Garcia L, Molina-Tijeras JA, Garcia F, Pischel I, Romero M, Duarte J, Diez-Echave P, Rodriguez-Cabezas ME, Rodriguez-Nogales A, Galvez J. The Antioxidant Activity of Thymus serpyllum Extract Protects against the Inflammatory State and Modulates Gut Dysbiosis in Diet-Induced Obesity in Mice. Antioxidants (Basel). 2022 May 28;11(6):1073. doi: 10.3390/antiox11061073. PMID 35739969
- [Background] Jaric S, Mitrovic M, Pavlovic P. Review of Ethnobotanical, Phytochemical, and Pharmacological Study of Thymus serpyllum L. Evid Based Complement Alternat Med. 2015;2015:101978. doi: 10.1155/2015/101978. Epub 2015 Jul 22. PMID 26265920
- [Background] Algieri F, Rodriguez-Nogales A, Garrido-Mesa N, Zorrilla P, Burkard N, Pischel I, Sievers H, Benedek B, Feistel B, Walbroel B, Rodriguez-Cabezas ME, Galvez J. Intestinal anti-inflammatory activity of the Serpylli herba extract in experimental models of rodent colitis. J Crohns Colitis. 2014 Aug;8(8):775-88. doi: 10.1016/j.crohns.2013.12.012. Epub 2014 Jan 8. PMID 24411672